CLINICAL TRIAL: NCT00554346
Title: A Randomized, Double Blind, Placebo-controlled Study to Assess the the Preemptive Benefit of Etoricoxib in Patients Receiving Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Ching-chuan Jiang, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200709062M
Record Dates: First submitted 2007-11-04; First posted 2007-11-06 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Post-operational Pain
Keywords: COX-2; post-operative ; sports injury; surgical pain
MeSH Terms: conditions — Athletic Injuries | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Etoricoxib 90mg
  Interventions: Drug: Arcoxia(etoricoxib 90 mg/tablet)
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Arcoxia(etoricoxib 90 mg/tablet)

INTERVENTIONS:
Drug: Arcoxia(etoricoxib 90 mg/tablet) — Arcoxia(etoricoxib 90 mg/tablet) or placebo, #1, 3 days

SUMMARY:
Post surgical pain associated with ligament reconstruction may persist for few days after the surgical procedure. Arcoxia is a new anti-inflammatory and analgesic drug that alleviate pain through oral administration. This study will test the safety and efficacy of Arcoxia in the management of post-operational pain in patients receive the ligament reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age ranged from 16~35 who have anterior cruciate ligament injury and/or associated injuries are scheduled for ACL reconstruction surgery.
2. Patient agrees to participate into this study and is willing to sign the patient informed consent form.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pain at rest at different timepoint after surgical procedures | From baseline(preoperation) to 3 days after

CONTACTS AND LOCATIONS:
Overall Officials: Ching Chuan Jiang, Professor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Alzheimer's Disease Education and Referral (ADEAR) Center — http://www.alzheimers.org